CLINICAL TRIAL: NCT04009629
Title: Dementia Risk and Dynamic Response to Exercise
Acronym: DYNAMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00142822; R21AG061548 (NIH)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease 2 Due to Apoe4 Isoform; Healthy Aging

STUDY DESIGN:
Intervention Model Description: Single visit, case-control study identified as an intervention due to the use of a single bout of aerobic exercise under NIH rules (grants.nih.gov/policy/clinical-trials/definition.htm)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise - apolipoprotein e4 carrier (Experimental): A single 15 minute bout of moderate intensity aerobic exercise for individuals with 1 or 2 copies of the APOE4 allele, the leading genetic risk factor for late-onset Alzheimer's dementia.
  Interventions: Behavioral: Moderate Intensity Aerobic Exercise
- Exercise - apolipoprotein e4 non-carrier (Experimental): A single 15 minute bout of moderate intensity aerobic exercise for individuals with 0 copies of the APOE4 allele, the leading genetic risk factor for late-onset Alzheimer's dementia.
  Interventions: Behavioral: Moderate Intensity Aerobic Exercise

INTERVENTIONS:
Behavioral: Moderate Intensity Aerobic Exercise — Participants will exercise for 15 minutes in a moderate age-predicted heart rate range. The study team will employ an exercise device such as a treadmill, cycle, or recumbent stepper to maintain control over workload.

SUMMARY:
Research suggests that physical exercise supports brain health and cognition as we age. The goal of this project is to examine the specific changes in brain blood flow and biological factors in the blood immediately after exercise in older adults who have the APOE4 gene, a genetic risk factor for developing Alzheimer's. Results from this study will help researchers and clinicians understand and measure changes in the body and brain as a function of exercise, and how those changes relate to Alzheimer's risk.

DETAILED DESCRIPTION:
The brain and cardiovascular system share common risk factors for age-related diseases such as hypertension, hypercholesterolemia, and genetics (e.g. APOE4). Because of this link, much work has focused on the role of cerebrovascular health in reducing dementia risk. Regular aerobic exercise has well-established benefits for cardiovascular health and has been repeatedly linked to better cognition, brain health, and lower risk of Alzheimer's disease (AD). Despite strong evidence for sustained cognitive and brain outcomes, the mechanisms relating aerobic exercise with brain health and cognition remain imprecisely defined. Amongst many potential mechanisms, cerebral blood flow (CBF) and blood-based biomarkers, such as neurotrophins, are promising targets for their shared association to brain and cardiovascular health. Prior investigations have largely attempted to measure change in these mechanisms under resting conditions after an extended exercise intervention with mixed and conflicting results. Further, studies have often not accounted for genetic differences that may blunt the effect of exercise. Unlike prior work, our innovative approach is to begin by characterizing the dynamic changes that result from an acute exercise challenge. A single bout of aerobic exercise temporarily increases CBF and prompts neurotrophin release. These transient changes ultimately drive long-term physiologic adaptation to exercise. Therefore, the study team will characterize the dynamic response to an acute, standardized bout of aerobic exercise in a group of nondemented older adults, comparing those who do and do not carry the APOE4 allele. The first aim will test if CBF response to an acute exercise challenge is blunted in APOE4 carriers. The second aim will similarly test the acute exercise response of blood-based biomarkers such as brain derived neurotrophic factor, insulin-like growth factor, and vascular endothelial growth factor in APOE4 carriers versus non-carriers. The study team expects that more accurately understanding the acute effects will provide valuable insight into how aerobic exercise supports cognitive function and brain health. Armed with this knowledge the field can optimize biomarker measurement for future exercise intervention randomized controlled trials, informing our long-term goal of identifying precision exercise prescription for AD prevention.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-85
* English speaking
* Normal or corrected hearing or vision,
* Without activity restrictions.

Exclusion Criteria:

* Clinically significant cognitive or psychiatric illness,
* Anti- coagulant use,
* High cardiovascular risk without physician clearance for exercise,
* Exercise-limiting musculoskeletal condition,
* MRI contraindications

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Vidoni, PT, PHD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Alzheimer's Disease Center, Fairway, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with unaffiliated investigators after completion of data collection and a reasonable amount of analysis and dissemination time. Contact the PI for further information.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Following a reasonable amount of analysis and dissemination time, the data will be available via request.
Access Criteria: Following institutional limits and recommendations and subject to use agreements.

REFERENCES:
- [Derived] Vidoni ED, Morris JK, Palmer JA, Li Y, White D, Kueck PJ, John CS, Honea RA, Lepping RJ, Lee P, Mahnken JD, Martin LE, Billinger SA. Dementia risk and dynamic response to exercise: A non-randomized clinical trial. PLoS One. 2022 Jul 8;17(7):e0265860. doi: 10.1371/journal.pone.0265860. eCollection 2022. PMID 35802628
- [Derived] White D, John CS, Kucera A, Truver B, Lepping RJ, Kueck PJ, Lee P, Martin L, Billinger SA, Burns JM, Morris JK, Vidoni ED. A methodology for an acute exercise clinical trial called dementia risk and dynamic response to exercise. Sci Rep. 2021 Jun 17;11(1):12776. doi: 10.1038/s41598-021-92177-0. PMID 34140586

RESULTS

PARTICIPANT FLOW:
Groups:
- APOE4 Carrier: Participants with 1 or 2 copies of the APOE4 allele, the leading genetic risk factor for late-onset Alzheimer's dementia.
- APOE4 Non-carrier: Participants with 0 copies of the APOE4 allele, the leading genetic risk factor for late-onset Alzheimer's dementia.
Period: Overall Study
Arm/Group | APOE4 Carrier | APOE4 Non-carrier
Started | 23 | 38
Completed | 21 | 38
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- APOE4 Carriers: Participants with 1 or 2 copies of the APOE4 allele, the leading genetic risk factor for late-onset Alzheimer's dementia.
- APOE4 Non-carriers: Participants with 0 copies of the APOE4 allele, the leading genetic risk factor for late-onset Alzheimer's dementia.
- Total: Total of all reporting groups
Arm/Group | APOE4 Carriers | APOE4 Non-carriers | Total
Number analyzed (Participants) | 23 | 38 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 23 | 38 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (5.1) | 73.3 (5.2) | 72.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 28 | 41
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 22 | 37 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 21 | 33 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 38 | 61

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Blood Flow Area Under Curve
Description: Cumulative cerebral blood flow measured by Arterial Spin Labeling MRI. The standard arterial spin labeling unit of measure is average milliliters per 100 grams of tissue per minute (mL/100g tissue/minute). For the present analysis, we summed perfusion over the entire acquisition period, 23.2 minutes, rather than averaging. Therefore the units are milliliters per 100 grams of tissue
Time Frame: ~24 minutes
Measure: Mean (Standard Deviation); unit: mL/100g tissue
Arm/Group | APOE4 Carrier | APOE4 Non-carrier
Number analyzed (Participants) | 21 | 38
mL/100g tissue | 715 (105.0) | 751 (87.6)

2. Secondary Outcome: Insulin-like Growth Factor-1 Change
Description: Change in circulating Insulin-like Growth Factor-1 from pre-to-post exercise
Time Frame: Pre-to-post intervention (~15 minutes)
Population: Blood collection failed on three individuals in the APOE4 carrier group. Outcome could not be analyzed.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | APOE4 Carrier | APOE4 Non-carrier
Number analyzed (Participants) | 20 | 38
picograms per milliliter | 2.25 (22.8) | 5.7 (27.8)

3. Secondary Outcome: Vascular Endothelial Growth Factor Change
Description: Change in circulating Vascular Endothelial Growth Factor from pre-to-post exercise
Time Frame: Pre-to-post intervention (~15 minutes)
Population: Blood collection failed on three individuals in the APOE4 carrier group. Outcome could not be analyzed.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Groups:
- APOE4 Non-carrier: Participants having zero copies of the APOE4 allele, the strongest late-onset genetic risk factor for Alzheimer's dementia.
Arm/Group | APOE4 Carrier | APOE4 Non-carrier
Number analyzed (Participants) | 20 | 38
picograms per milliliter | -1.01 (10.6) | 1.83 (11.1)

4. Secondary Outcome: Brain Derived Neurotrophic Factor Change
Description: Change in circulating Brain Derived Neurotrophic Factor from pre-to-post exercise
Time Frame: Pre-to-post intervention (~15 minutes)
Population: Blood collection failed on three individuals in the APOE4 carrier group. Outcome could not be analyzed.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | APOE4 Carrier | APOE4 Non-carrier
Number analyzed (Participants) | 20 | 38
picograms per milliliter | -219 (641) | 208 (706)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Adverse events were defined as any untoward or unfavorable medical occurrence in a human subject participant, including any abnormal sign, symptom, or disease, temporally associated with the participants' involvement in the research, whether or not considered related to participation in the research.
Arm/Group | APOE4 Carrier | APOE4 Non-carrier
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/38
Other Adverse Events (participants affected / at risk) | 1/23 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APOE4 Carrier (N=23) | APOE4 Non-carrier (N=38)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT04009629/Prot_SAP_000.pdf